CLINICAL TRIAL: NCT03688178
Title: DC Migration Study to Evaluate TReg Depletion In GBM Patients With and Without Varlilumab
Acronym: DERIVe
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Annick Desjardins, MD (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, MD, Assistant Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00082570
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Dendritic cells; Temozolomide; Duke University; Varlilumab; Desjardins
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; varlilumab; Toxoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Assignment to Groups 1 and 2 is blinded, and neither the study team nor the subject knows which pre-conditioning regimen is given. Assignment to Group 3 is not blinded, and the subject and study team know that Td preconditioning and Varlilumab is given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gr1: DC vaccine (DC pre-conditioning) (Experimental): Patients will receive TMZ at a target dose of 150-200 mg/m^2/d for 5 days every 4 (+2) weeks for up to 12 cycles. DC vaccines will be administered in equal amounts to both inguinal regions. DC vaccines #1-3 occur every 2 weeks and all subsequent vaccines (up to 10) occur monthly. Group 1 patients will receive autologous unpulsed DC vaccines administered to a single side of the groin and saline administered to the contralateral side the day prior to the 4th DC vaccine as pre-conditioning.
  Interventions: Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs; Drug: Temozolomide; Biological: Unpulsed DCs
- Gr2: DC Vaccine (Td pre-conditioning) (Experimental): Patients will receive TMZ at a target dose of 150-200 mg/m^2/d for 5 days every 4 (+2) weeks for up to 12 cycles. DC vaccines will be administered in equal amounts to both inguinal regions. DC vaccines #1-3 occur every 2 weeks and all subsequent vaccines (up to 10) occur monthly. Group 2 patients will receive a single dose of Td toxoid administered to a single side of the groin and saline administered to the contralateral side the day prior to the 4th DC vaccine, which is always given bilaterally at the groin site.
  Interventions: Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs; Drug: Temozolomide; Biological: Td
- Gr3:DC Vaccine+varlilumab(Td pre-conditioning) (Experimental): Patients will receive TMZ at a target dose of 150-200 mg/m^2/d for 5 days every 4 (+2) weeks for up to 12 cycles. DC vaccines will be administered in equal amounts to both inguinal regions. DC vaccines #1-3 occur every 2 weeks and all subsequent vaccines (up to 10) occur monthly. Group 3 patients will receive the first 3 DC vaccines every 2 weeks, same as Groups 1 and 2, but they will also receive varlilumab intraveneously (IV) 7 days before vaccine #1 and again at the same visit as vaccine #1, as well as 7 days before every DC vaccine except vaccine #2. Prior to the 4th vaccine, patients will receive a single dose of Td toxoid administered to a single side of the groin and saline administered to the contralateral side.
  Interventions: Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs; Drug: Temozolomide; Biological: Varlilumab; Biological: Td

INTERVENTIONS:
Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs — 2x10^7 human CMV pp65-LAMP mRNA-pulsed autologous DCs are given intradermally and bilaterally at the groin site (divided equally to both inguinal regions). Patients will receive up to a total of 10 DC vaccines.
Drug: Temozolomide — Temozolomide is a standard chemotherapy given to all enrolled patients at a targeted dose of 150-200mg/m2/d for 5 days every 4 (+ 2) weeks for up to 12 cycles (patients with unmethylated MGMT gene promoter will receive only cycle 1)
  Other Names: Temodar; TMZ; Temodal
Biological: Varlilumab — Varlilumab is an agonist anti-CD27 monoclonal antibody
  Other Names: anti-CD27
  Arms: Gr3:DC Vaccine+varlilumab(Td pre-conditioning)
Biological: Td — A single dose of Td toxoid (1 flocculation unit, Lf, in 0.4 mLs) administered to a single side of the groin given intradermally
  Other Names: Tetanus-diphtheria (Td) toxoid; Td pre-conditioning
  Arms: Gr2: DC Vaccine (Td pre-conditioning); Gr3:DC Vaccine+varlilumab(Td pre-conditioning)
Biological: Unpulsed DCs — Patients in Group I will receive 1 x 10^6 autologous unpulsed DCs in saline administered to a single side of the groin intradermally 1 day before the fourth vaccine.
  Other Names: Unpulsed DCs pre-conditioning
  Arms: Gr1: DC vaccine (DC pre-conditioning)

SUMMARY:
Patients with newly diagnosed glioblastoma will be consented following tumor resection then undergo leukapheresis for harvest of peripheral blood leukocytes for generation of dendritic cells. Subjects will then receive standard of care (planned 6 weeks) radiation therapy (RT) and concurrent temozolomide (TMZ) at a standard targeted dose of 75 mg/m2/day.

The study cycle of TMZ comprises a targeted dose of 150-200mg/m2/day for 5 days every 4 (+2) weeks for up to 12 cycles (patients with unmethylated MGMT gene promoter will receive only cycle 1). All patients will receive up to a total of 10 DC vaccines called pp65 CMV dendritic cells (DC). Dendritic Cell (DC) vaccines #1-3 will be given every two weeks, thus delaying the initiation of TMZ cycle 2 for patients receiving TMZ. All remaining TMZ/vaccine cycles will be 4 (+2) weeks in length.

After the first 3 DC vaccines given during Cycle 1 of TMZ, the remaining DC vaccine injections are given on Day 21 (+/- 2 days) of each TMZ cycle. Subjects with unmethylated MGMT will only receive one cycle of adjuvant TMZ; however, their vaccine schedule will follow the same 4 (+ 2) week TMZ cycle schedule.

Following RT, patients will be randomized into 1 of 3 groups. Groups 1 and 2 will be blinded. The groups differ in the type of pre-conditioning received prior to DC vaccine #4; additionally, Group 3 will be receiving infusions of varlilumab 7 days prior to and with vaccine #1 and 7 days prior to vaccine #3+. The pre-conditioning for each group is as follows: Group 1: Unpulsed DC pre-conditioning prior to DC vaccine #4; Group 2: Tetanus-diphtheria (Td) pre-conditioning prior to DC vaccine #4; Group 3: Td pre-conditioning prior to DC vaccine #4 and varlilumab infusion at 7 days prior to each DC vaccine (except DC vaccine #2) with Td pre-conditioning prior to vaccine #4.

DETAILED DESCRIPTION:
Human cytomegalovirus (CMV) is a common endemic β-Herpesvirus, and over half of adults have been infected with CMV. CMV does not usually cause significant clinical disease but can cause health problems for people with weakened immune systems. Expression of proteins unique to human CMV has been reported within a large proportion of malignant gliomas (MGs), including detection of the human CMV immunodominant protein pp65-LAMP (pp65-lysosomal-associated membrane protein). Human CMV antigens were not detected in surrounding normal brain samples. The presence of highly-immunogenic human CMV antigens within MGs affords a unique opportunity to target these tumors immunologically.

Dendritic cells (DCs) are antigen-presenting cells in the immune system. DCs are activated then migrate to the lymph nodes to interact with T cells and B cells, which initiates the adaptive immune response. This study generates autologous DCs from peripheral blood leukocytes obtained from the subject during leukapheresis. RNA transfection is the method used in this study for loading antigens onto DCs. DCs are pulsed with human CMV pp65-LAMP mRNA.

Tetanus-diphtheria (Td) toxoid is used for active immunization in children and adults against infection with the bacteria Clostridium tetani and Corynebacterium diphtheria. It is thought that Td toxoid induces an inflammatory milieu within the intradermal vaccine site, thereby promoting the migration of injected tumor-specific DCs. Additionally, in the context of vaccinating the host with tumor-derived peptides, conditioning the vaccine site with Td toxoid has demonstrated enhanced immunogenicity with these peptides. Previous trials have suggested that giving the Td prior to immunotherapy may help improve the effectiveness of the DC vaccine by activating the immune response. This study will further examine whether Td helps activate the immune response by comparing subjects who receive Td pre-conditioning to subjects who receive autologous unpulsed DCs as pre-conditioning.

Varlilumab is a fully human monoclonal antibody (mAb) that targets CD27, a critical molecule in the activation pathway of lymphocytes. Varlilumab is an agonist anti-CD27 mAb that has been shown to activate human T cells in the context of T cell receptor stimulation. In pre-clinical models, varlilumab has been shown to mediate anti-tumor effects and may be particularly effective in combination with other immunotherapies. Anti-CD27 mAb has emerged as a novel costimulatory immune modulator that depletes TRegs without impairing activated effector T cells to improve antitumor immunity. We hypothesize that TReg inhibition through Varlilumab may increase polyfunctional immune responses to CMV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age.
* Glioblastoma with definitive resection prior to enrollment, with residual radiographic contrast enhancing disease on the post-operative CT or MRI of <1 cm in maximal diameter in any plane.
* Able to receive SOC RT/TMZ for approximately 6 weeks duration and of more than 54GY
* MRI post RT does not show progressive disease outside the radiation field
* Enough tumor tissue available for determination of MGMT gene promoter status.
* CMV Seropositive
* KPS of ≥ 70%
* Hemoglobin ≥ 9.0 g/dl, ANC ≥ 1,000 cells/µl, platelets ≥ 100,000 cells/µl.
* Serum creatinine ≤3 times institutional upper limit of normal for age, serum SGOT ≤ 3 times institutional upper limit of normal f.or age and bilirubin ≤ 1.5 times upper limit of normal prior to starting TMZ cycle 1 (Exception to bilirubin criteria: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3 x ULN is acceptable).
* Signed informed consent approved by the Institutional Review Board.
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [IUD; only hormonal], sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to first study treatment.
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drugs.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* Patients with known potentially anaphylactic allergic reactions to gadolinium-DTPA.
* Patients who cannot undergo MRI due to obesity or to having certain metal in their bodies (specifically pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates).
* Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, radiological evidence of multifocal disease, or leptomeningeal disease.
* Severe, active comorbidity, including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization;
  * Transmural myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study initiation;
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy;
  * Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
  * Known HIV and Hepatitis C positive status;
  * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy;
  * Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin. (Treatment with tamoxifen or aromatase inhibitors or other hormonal therapy that may be indicated in prevention of prior cancer disease recurrence, are not considered current active treatment.)
* Patients are not permitted to have had any other conventional therapeutic intervention other than steroids prior to enrollment outside of standard of care chemotherapy and radiation therapy. Patients who receive previous inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies will be excluded.
* Current, recent (within 4 weeks of the administration of this study agent), or planned participation in an experimental drug study.
* Known history of autoimmune disease (with the exceptions of medically-controlled hypothyroidism and Type I Diabetes Mellitus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Median Overall Survival (OS) of Subjects Receiving Td pre-conditioning | 5 years
  OS is defined as the time in months between randomization and death, or last follow-up if alive (Groups 1 and 2). Kaplan-Meier methods will be used to estimate median OS
Safety of administering Varlilumab to GBM patients receiving temozolomide and dendritic cell vaccines ± Td pre-conditioning as measured by the percentage of patients with unacceptable toxicity regardless of attribution | 5 years
  Percentage of patients with unacceptable toxicity (all Groups)
Median percent change between baseline, assessed on day 14, and nadir levels of Treg before the time that the second cycle of adjuvant TMZ would be administered. Treg determined by flow cytometry (CD3+ CD4+ CD25+ Foxp3+). | 50 days
  Change between baseline and nadir before the 2nd cycle of TMZ (Combined Groups 1 and 2, Group 3)

SECONDARY OUTCOMES:
Median Overall Survival (OS) of Subjects Receiving DC vaccines, varlilumab, and Td pre-conditioning | 5 years
  OS is defined as the time in months between randomization and death, or last follow-up if alive (Group 3). Kaplan-Meier methods will be used to estimate median OS
Median Progression-free Survival (PFS) | 5 years
  PFS is defined as the time between randomization and initial failure (disease progression or death) (all Groups). If the patient remains alive without disease progression, PFS will be censored at the time of last follow-up. Kaplan-Meier methods will be used to estimate median PFS
Median Chemokine (C-C motif) ligand 3 (CCL3) Levels in Serum at 24, 48, and 72 hours after Pre-conditioning | 2 days
  CCL3 levels in serum 24, 48, and 72 hours after pre-conditioning by multiplex. The median CCL3 level will be presented

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/

DOCUMENTS (1):
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03688178/ICF_001.pdf